CLINICAL TRIAL: NCT05291728
Title: Screening for Early Gastric Cancer in Shaanxi Province
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021036
Record Dates: First submitted 2022-02-24; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: Early Gastric Cancer
Keywords: early GC,Hp infection,FD, GERD , precancerous lesions
MeSH Terms: conditions — Stomach Neoplasms; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study collect the relevant data of local residents over 20 years old in 11 regions of Shaanxi Province, The basic information of the subjects was collected by filling in the questionnaire, and serum helicobacter pylori antibody detection was completed at the same time. The expert group determined the high-risk population of gastric cancer after comprehensive evaluation. All the high-risk population of gastric cancer without contraindications underwent electronic gastroscopy in the designated hospital after signing the informed consent. By collecting and analyzing data, early gastric cancer screening was completed and a new gastric cancer risk assessment model was established to evaluate the prevalence of dyspepsia, gastroesophageal reflux disease and precancerous lesions in the natural population of Shaanxi Province, as well as helicobacter pylori infection, radical treatment and recurrence rate.

DETAILED DESCRIPTION:
From October 2020 to October 2026, after obtaining the informed consent of local residents over 20 years old in 11 regions of Shaanxi Province, the subjects' social demographic characteristics, living and eating habits, and previous diseases were collected by filling in questionnaires, and serum helicobacter pylori antibody was detected at the same time. After comprehensive assessment by the expert group, the high-risk population of gastric cancer was determined. All high-risk population of gastric cancer without contraindications underwent electronic gastroscopy in designated hospitals after signing informed consent. By collecting and analyzing data, early gastric cancer screening was completed and a new gastric cancer risk assessment model was established to evaluate the prevalence of dyspepsia, gastroesophageal reflux disease and precancerous lesions in the natural population of Shaanxi Province, as well as helicobacter pylori infection, radical treatment and recurrence rate. In this project, the research group was responsible for formulating the plan, designing the questionnaire, and conducting quality control and grass-roots guidance tour. Guanghua Science and Technology Foundation provided public welfare assistance, and distributed and collected questionnaires with the assistance of grass-roots clinics. Finally, the research group sorted out and analyzed the data.

ELIGIBILITY:
Inclusion Criteria:

* Local resident over 20 years old.
* Obtain verbal informed consent of the subject.

Exclusion Criteria:

* Refused to participate in this research project.
* Questionnaires or serological tests for helicobacter pylori antibodies were not completed.
* This study was not completed due to other reasons.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be carried out in 11 regions of Shaanxi Province from October 2020 to October 2026. Data of permanent resident population (registered population combined with floating population) in the region will be obtained by the local government, and all permanent residents over 20 years old in each region will be identified as the target population. It is preliminarily estimated that the permanent residents over 20 years old in each region of Shaanxi account for about 20%-60% of the total population, and the screening target of permanent residents over 20 years old in each region is finally established in this project.
Sampling Method: Probability Sample
Enrollment: 12500000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
the detection rate of early gastric cancer | 2020.10.01-2026.10.01
  Patients at high risk of gastric cancer were assessed by questionnaire and Hp test results, and then underwent gastroscopy.Then analyse the detection rate of early gastric cancer.

SECONDARY OUTCOMES:
the prevalence of dyspepsia, gastroesophageal reflux disease and precancerous lesions in the natural population of Shaanxi Province, as well as the prevalence of helicobacter pylori infection, radical treatment and recurrence rate. | 2020.10.01-2026.10.01
  Basic information, Hp antibody detection results and gastroscopy results were collected,and then analyse the prevalence of dyspepsia, gastroesophageal reflux disease and precancerous lesions in the natural population of Shaanxi Province, as well as the prevalence of helicobacter pylori infection, radical treatment and recurrence rate.

CONTACTS AND LOCATIONS:
Overall Officials: jinhai Wang, MD, Study Director — Second Affilated Hospital of Xi'an Jiaotong University
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No